CLINICAL TRIAL: NCT00705913
Title: A Randomized Study to Compare Sizing, Implant Techniques and Hemodynamic Performance Between the Mitroflow and the Carpentier-Edwards Magna Pericardial Tissue Valves in the Aortic Position
Brief Title: Randomized Sizing and Hemodynamic Study Mitroflow vs. Magna
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRVSS-02
Record Dates: First submitted 2008-06-18; First posted 2008-06-27 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-11

CONDITIONS: Aortic Valve Disease
Keywords: aortic valve; heart valve; valve replacement; valve disease
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mitroflow Aortic Pericardial Heart Valve (CarboMedics)
  Interventions: Device: Mitroflow Aortic Pericardial Heart Valve (CarboMedics)
- 2 (Active Comparator)
  Interventions: Device: Carpentier-Edwards Magna Tissue Valve

INTERVENTIONS:
Device: Mitroflow Aortic Pericardial Heart Valve (CarboMedics) — Study to compare sizing, implant techniques and hemodynamics of the Mitroflow Pericardial valve as compared to the Edwards Magna valve
  Arms: 1
Device: Carpentier-Edwards Magna Tissue Valve — Study to compare sizing, implant techniques and hemodynamics of the Mitroflow Valve as compared to the Edwards Magna valve
  Arms: 2

SUMMARY:
The purpose of this study is to compare sizing,implant techniques, and hemodynamics between the Mitroflow Pericardial Aortic Valve and the Edwards Magna Heart Valve.

DETAILED DESCRIPTION:
Comparisons of valve types are often made according to labeled valve sizes. There is growing evidence that in the majority of cases the actual sizer and valve dimensions vary from the labeled diameters, which may not be related to any hemodynamically meaningful dimension. The disagreement between the true valve dimensions and the labeled valve size may render comparisons based on labeled size meaningless

ELIGIBILITY:
Inclusion Criteria:

* Patients who are indicated for implant with a bioprosthetic valve in the aortic position according to the current practice for valve selection at the center.

Exclusion Criteria:

* Less than 18 years of age
* Emergency Surgery
* Pre-existing valve prothesis in the aortic position
* Aortic root replacements or enlargements
* Active endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2008-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Determine which of the two valve types, the Mitroflow or Magna valve, will demonstrate lower pressure gradients relative to aortic annulus | 6 months

SECONDARY OUTCOMES:
Determine which of the two valve types, the Mitroflow or Magna valve, will demonstrate higher ratio of EOA to the aortic annulus area. | 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - Sharp Memorial Hospital, San Diego, California
  - Pepin Heart Hospital, Tampa, Florida
  - St. Luke's Medical Center, Kansas City, Kansas
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - St. John's Medical Research Inst., Springfield, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - The Ohio State University Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Heart Hospital Baylor Plano, Plano, Texas
- Canada (2):
  - St.Boniface General Hospital, Winnipeg, Manitoba
  - Hopital Laval, Sainte-Foy, Quebec